CLINICAL TRIAL: NCT04660201
Title: A Phase 1, Randomized, Parallel-Group, Double-Blind Trial of AV7909 (Liquid) and Thermostable AV7909 (Lyophilized) in Healthy Adult Volunteers
Brief Title: Anthrax AV7909 Liquid vs Lyophilized
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-0093
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2020-09

CONDITIONS: Anthrax; Anthrax Immunisation
Keywords: Anthrax; AV7909 (Liquid); Healthy Adult Volunteers; Immunogenicity; Phase 1; Safety; Thermostable AV7909 (Lyophilized); Vaccine
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): AV7909 liquid formulation will be administered 0.5mL intramuscularly in a 2-dose schedule, 2 weeks apart (on Day 1 and Day 15). N=20
  Interventions: Biological: AV7909
- Group 2 (Active Comparator): AV7909 lyophilized formulation will be administered 0.5mL intramuscularly in a 2-dose schedule, 2 weeks apart (on Day 1 and Day 15). N=20
  Interventions: Biological: AV7909

INTERVENTIONS:
Biological: AV7909 — AV7909 (Liquid Formulation) is an investigational vaccine that is a preformulated, sterile, milky-white suspension for IM injection. It consists of the Anthrax Vaccine Adsorbed (AVA) bulk drug substance and CPG 7909 adjuvant
  Arms: Group 1
Biological: AV7909 — AV7909 (Lyophilized Formulation) is a thermostable, lyophilized version of the liquid AV7909 formulation. Sterile, milky-white suspension for intramuscular injection. It consists of polysorbate 80, CPG7909 adjuvant and AVA bulk drug substance
  Arms: Group 2

SUMMARY:
This is a randomized, parallel-group, double-blind, Phase 1 study designed to assess safety, tolerability and immunogenicity 2 formulations of adjuvanted anthrax vaccine (AV7909), lyophilized and liquid. Forty healthy young adults, 18 to 45 years old, inclusive, who meet all eligibility criteria, will be randomly allocated to one of two study groups in a 1:1 ratio: 20 will receive AV7909 as the thermostable lyophilized product and 20 will receive AV7909 as the liquid product. The vaccines will be given intramuscularly in a 2-dose schedule, 2 weeks apart.

Safety will be assessed by evaluation of non-serious unsolicited Adverse Events, Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs) [the AESIs collected in this study are Potentially Immune-Mediated Medical Conditions (PIMMCs)], and by laboratory evaluations. Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions in the week after each study vaccination.

Immunogenicity testing will include performing serological assays to assess for toxin neutralizing antibodies (reported as ED50 and NF50), the gold standard assay for assessing response and protection following anthrax vaccines, prior to vaccination and on approximately Days 8, 15, 22, 29, 64, 195, and 380. In addition, anti-PA IgG antibodies will be measured by ELISA from the serum of participants, on those same days. The primary safety objective of this study is to assess the safety of lyophilized and liquid formulations of AV7909. The primary tolerability objective is to assess the tolerability of lyophilized and liquid formulations of AV7909.

DETAILED DESCRIPTION:
This is a randomized, parallel-group, double-blind, Phase 1 study designed to assess safety, tolerability and immunogenicity of 2 formulations of adjuvanted anthrax vaccine (AV7909), lyophilized and liquid. Forty healthy young adults, 18 to 45 years old, inclusive, who meet all eligibility criteria, will be randomly allocated to one of two study groups in a 1:1 ratio: 20 will receive AV7909 as the thermostable lyophilized product and 20 will receive AV7909 as the liquid product. Stratification by age category and by gender will assure that near equal numbers of younger (18-30 years) and older (31-45 years) males and females are assigned to each vaccine. The vaccines will be given intramuscularly in a 2-dose schedule, 2 weeks apart.

Safety will be assessed by evaluation of non-serious unsolicited Adverse Events, Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs) [the AESIs collected in this study are Potentially Immune-Mediated Medical Conditions (PIMMCs)], and by laboratory evaluations. Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions in the week after each study vaccination.

Immunogenicity testing will include performing serological assays to assess for toxin neutralizing antibodies (reported as ED50 and NF50), the gold standard assay for assessing response and protection following anthrax vaccines, prior to vaccination and on approximately Days 8, 15, 22, 29, 64, 195, and 380. In addition, anti-PA IgG antibodies will be measured by ELISA from the serum of participants, on those same days. The primary safety objective of this study is to assess the safety of lyophilized and liquid formulations of AV7909. The primary tolerability objective is to assess the tolerability of lyophilized and liquid formulations of AV7909. The secondary immunogenicity objective of this study is to obtain initial estimate of comparative immunogenicity of liquid and lyophilized formulations of AV7909.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Understand and comply with planned study procedures, including completion of the electronic memory aid, and be available for all study visits.
3. Agree to the collection of venous blood, per protocol.
4. Have adequate venous access for phlebotomies.
5. Be a male or non-pregnant female, 18 to 45 years of age, inclusive, at the time of enrollment.
6. Be in good health.*

   * As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, which would affect the assessment of the safety of participants or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, should be stable (not worsening) for the last 60 days (no hospitalizations, emergency room or urgent care for condition, or invasive medical procedure and no adverse symptoms that need medical intervention such as medication change indicative of worsening/supplemental oxygen). This includes no change in chronic prescription medication, dose or frequency, indicative of worsening disease, in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening or treatment of continued symptoms of medical diagnosis or condition. Herbals, vitamins, and supplements are permitted.
7. Have an oral temperature less than 100.0 degrees Fahrenheit.
8. Have a pulse 51 to 100 beats per minute, inclusive.
9. Have a systolic blood pressure 85 to 140 mmHg, inclusive.
10. Have a diastolic blood pressure 55 to 90 mmHg, inclusive.
11. Have a calculated body mass index (BMI) less than or equal to 35.0 kg/m2 at screening.
12. Screening laboratories are within acceptable parameters:

    * BUN <23 mg/dL
    * Serum creatinine (female) <1.3 mg/dL
    * Serum creatinine (male) < 1.4 mg/dL
    * Alkaline phosphatase (female) <147 U/L
    * Alkaline phosphatase (male) <192 U/L
    * ALT (aka SGPT) <68 U/L
    * Total bilirubin < 1.3 mg/dL
    * Hemoglobin (female) >10.9 g/dL
    * Hemoglobin (male) > 12.4 g/dL
    * White blood cell count 3000-12,000 cells/mm3
    * Absolute eosinophil count <1201 cells/mm3
    * Absolute neutrophil count >1200 cells/mm3
    * Platelets >126,000 cells/mm3
    * Hemoglobin A1C <6.5%
    * Urine for Drugs of Abuse (amphetamines, barbiturates, benzodiazepines, cocaine, methadone, opiates, oxycodone/oxymorphone, phencyclidine (PCP), and propoxyphene). All negative
    * HBsAg Non-reactive
    * HCV antibodies Negative
    * HIV 4th generation test Negative
13. Have no clinically significant findings on 12-lead electrocardiogram.*

    * Clinical significance will be determined by a cardiologist. Examples of findings that will lead to exclusion are significant left ventricular hypertrophy, right or left bundle branch block, advanced A-V heart block, non-sinus rhythm (excluding isolated premature atrial contractions), pathologic Q wave abnormalities, significant ST-T wave changes, prolonged QTc interval.
14. Heterosexually active females of childbearing potential* must use an acceptable contraception method** from at least 30 days before the first until 60 days after the second study vaccination.

    * Not sterilized via bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses, if menopausal.

      * Includes full abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more or shown to be azoospermic prior to the participant receiving the study vaccination, barrier methods such as condoms or diaphragms/cervical cap, intrauterine devices, NuvaRing(R), tubal ligation, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
15. Females of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.
16. For a female with potential to become pregnant, she understands that in the event of pregnancy during the study she will be asked to allow us to follow her during pregnancy through outcome.
17. Must agree to have blood collected, stored, and potentially used for auto-antibody studies (if a suspected Potentially Immune-Mediated Medical Conditions (PIMMC) occurs in this participant).

Exclusion Criteria:

1. Have an acute illness*, as determined by the site principal investigator (PI) or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters and systemic reactogenicity events as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation.*

   *Including acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.*

   *These include oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination, or high-dose inhaled corticosteroids within 30 days prior to study vaccination, with high-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE. Intranasal corticosteroids are not exclusionary. Low and moderate potency topical corticosteroids are permitted.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy. Non-melanoma treated skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), chronic hepatitis B, or hepatitis C infection.
7. Have known hypersensitivity or allergy to any components of the study vaccines (Anthrax Vaccine Adsorbed (AVA), CPG adjuvants, aluminum, benzethonium chloride [phemerol], formaldehyde).
8. Have a history of receipt or plan to receive, while enrolled in this study, a licensed or unlicensed anthrax vaccine (except for the vaccines under study herein).
9. Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).*

   *Adverse Events of Special Interest
10. Have a history of alcohol or drug abuse within 5 years prior to study enrollment or test positive on the screening urine test for drugs of abuse.
11. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere* with participant compliance or safety evaluations.

    *As determined by the site PI or appropriate sub-investigator.
12. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
13. Received or plan to receive a licensed, live vaccine within 30 days before or after each study vaccination.
14. Received or plan to receive a licensed, inactivated vaccine within 14 days before or after each study vaccination.
15. Have a known history of documented anthrax disease or suspected exposure to anthrax.
16. Received immunoglobulin or other blood products, except Rho(D) immunoglobulin, within 90 days prior to study vaccination.
17. Received an experimental agent* within 30 days prior to the study vaccination or expect to receive another experimental agent** during the trial-reporting period.***

    * Including vaccine, drug, biologic, device, blood product, or medication.

      * Other than from participation in this trial. ***Approximately 12 months after the second study vaccination.
18. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the trial-reporting period.**

    *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

    **Approximately 12 months after the second study vaccination.
19. Female participants who are breastfeeding or plan to breastfeed from the time of the first study vaccination through 30 days after the second study vaccination.
20. Planning to donate blood within 4 months following second vaccination.
21. Planned elective surgery during study participation.
22. Member or immediate family member of the site research staff found on the delegation log.
23. Previously served in the military any time after 1990 and/or plan to enlist in the military at any time during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females, 18 to 45 years of age, inclusive, who met all eligibility criteria. They were recruited from the general population at the participating site: University of Maryland, Baltimore. Participants were enrolled between 25May2022 and 09Sep2022.
Groups:
- Liquid AV7909: AV7909 liquid product administered intramuscularly in a 2-dose schedule, 2 weeks apart (Day 1 and Day 15).
  AV7909 is an investigational vaccine manufactured by Emergent BioSolutions (Emergent) combining the currently licensed Anthrax Vaccine Adsorbed (AVA) with the adjuvant CPG 7909. CPG 7909 is a lyophilized powder manufactured by Avecia Nitto Denko in Milford, MA. CPG 7909's natural deoxyribonucleic acid phosphodiester backbone has been modified to a phosphorothioate backbone, providing the molecule with increased stability and resistance to degradation for improved in vivo activity.
  Liquid AV7909 is a preformulated, sterile, milky-white suspension (when mixed) for intramuscular injection.
- Lyophilized AV7909: AV7909 thermostable lyophilized product administered intramuscularly in a 2-dose schedule, 2 weeks apart (Day 1 and Day 15).
  AV7909 is an investigational vaccine manufactured by Emergent BioSolutions (Emergent) combining the currently licensed Anthrax Vaccine Adsorbed (AVA) with the adjuvant CPG 7909. CPG 7909 is a lyophilized powder manufactured by Avecia Nitto Denko in Milford, MA. CPG 7909's natural deoxyribonucleic acid phosphodiester backbone has been modified to a phosphorothioate backbone, providing the molecule with increased stability and resistance to degradation for improved in vivo activity.
  Thermostable AV7909 is a lyophilized version of the liquid AV7909 formulation which, after reconstitution, is a sterile, milky-white suspension for intramuscular injection. The Thermostable AV7909 Bulk Intermediate Product is manufactured at Emergent's Baltimore, MD facility by addition of Polysorbate 80 and CPG7909 adjuvant to AVA Bulk Drug Substance produced by Emergent's Manufacturing facility at Lansing, MI. The Thermostable AV7909 Final Drug Product is manufactured by Integrity Bio Inc.
  The AV7909 lyophilized product is mixed with a diluent of United States Pharmacopeia (USP) grade Sterile Water For Injection provided by Fisher BioServices.
Period: Overall Study
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received the first dose of study vaccine.
Groups:
- Liquid AV7909: AV7909 liquid product administered intramuscularly in a 2-dose schedule, 2 weeks apart (Day 1 and Day 15).
- Lyophilized AV7909: AV7909 thermostable lyophilized product administered intramuscularly in a 2-dose schedule, 2 weeks apart (Day 1 and Day 15).
- Total: Total of all reporting groups
Arm/Group | Liquid AV7909 | Lyophilized AV7909 | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.7) | 29.8 (5.1) | 29.3 (5.4)
Age, Customized [Count of Participants; unit: Participants]
  18-30 years old | 13 | 12 | 25
  31-45 years old | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 17 | 31
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
Height [Mean (Standard Deviation); unit: cm] | 170.40 (9.36) | 172.09 (9.22) | 171.22 (9.21)
Weight [Mean (Standard Deviation); unit: kg] | 75.79 (17.67) | 75.43 (15.65) | 75.61 (16.51)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.87 (4.47) | 25.31 (3.88) | 25.60 (4.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) included any AE or suspected adverse reaction that, in the view of either the site PI (or appropriate sub-investigator) or sponsor, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, was a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, was a congenital anomaly/birth defect, or may have jeopardized the participant and required medical or surgical intervention to prevent one of the aforementioned outcomes.
Time Frame: Day 1 through Day 380
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Clinical Safety Laboratory Adverse Events (AEs).
Description: Clinical safety laboratory parameters include blood urea nitrogen (BUN), serum creatinine, alkaline phosphatase, alanine aminotransferase (ALT), total bilirubin, hemoglobin, hemoglobin decrease from baseline, white blood cell (WBC) count, absolute eosinophil count, absolute neutrophil count, platelets, aspartate aminotransferase (AST), random glucose, urine protein, and urine glucose.
Time Frame: Day 29
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants
  Blood urea nitrogen (BUN) | 0 | 0
  Creatinine | 0 | 1
  Alkaline phosphatase (ALP) | 0 | 0
  Alanine aminotransferase (ALT) | 0 | 0
  Total bilirubin | 1 | 0
  Hemoglobin | 1 | 0
  Hemoglobin decrease from baseline | 3 | 5
  White blood cell (WBC) count | 0 | 0
  Absolute eosinophil count | 0 | 0
  Absolute neutrophil count | 0 | 0
  Platelets: number analyzed (Participants) | 21 | 19
  Platelets | 0 | 0
  Aspartate aminotransferase (AST): number analyzed (Participants) | 4 | 5
  Aspartate aminotransferase (AST) | 0 | 0
  Random glucose: number analyzed (Participants) | 4 | 5
  Random glucose | 0 | 1
  Urine protein: number analyzed (Participants) | 4 | 5
  Urine protein | 1 | 0
  Urine glucose: number analyzed (Participants) | 4 | 5
  Urine glucose | 0 | 0

3. Primary Outcome: Number of Participants With Protocol-specified Adverse Events of Special Interest (AESIs)
Description: Adverse events of special interest (AESIs) in this study were potentially immune-mediated medical conditions (PIMMCs). A list of PIMMCs was provided in the study protocol, including gastrointestinal disorders, liver disorders, metabolic diseases, musculoskeletal disorders, neuroinflammatory disorders, skin disorders, vasculitides, and autoimmune syndromes.
Time Frame: Day 1 through Day 380
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs).
Description: Adverse events (AEs) characterized by unscheduled medical attention, defined as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason, were designated as medically attended adverse events (MAAEs).
Time Frame: Day 1 through Day 380
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants | 9 | 8

5. Primary Outcome: Number of Participants With Unsolicited, Non-serious Adverse Events (AEs).
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. The occurrence of an unsolicited AE may have come to the attention of study personnel during study visits and interviews for medical care, or upon review by a study monitor.
Time Frame: Day 1 through Day 64
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants | 14 | 13

6. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactogenicity Events Following First Study Vaccination.
Description: Injection site and systemic reactogenicity events were solicited daily throughout the week following each study vaccination. The number of participants reporting each event on any day following first vaccination is presented. Injection site reactogenicity events included pruritus, ecchymosis, erythema, edema/induration, pain, and tenderness. Systemic reactogenicity events included fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea.
Time Frame: Day 1 through Day 8
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants
  Pain | 19 | 12
  Tenderness | 19 | 20
  Pruritus | 2 | 2
  Ecchymosis (functional grade) | 2 | 2
  Ecchymosis (measurement grade) | 2 | 2
  Erythema (functional grade) | 0 | 2
  Erythema (measurement grade) | 0 | 2
  Edema/Induration (functional grade) | 2 | 2
  Edema/Induration (measurement grade) | 1 | 1
  Fever | 1 | 2
  Feverishness | 5 | 5
  Fatigue | 16 | 13
  Malaise | 10 | 4
  Myalgia | 11 | 6
  Arthralgia | 5 | 2
  Headache | 10 | 13
  Nausea | 4 | 3

7. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactogenicity Events Following Second Study Vaccination.
Description: Injection site and systemic reactogenicity events were solicited daily throughout the week following each study vaccination. The number of participants reporting each event on any day following second vaccination is presented. Injection site reactogenicity events included pruritus, ecchymosis, erythema, edema/induration, pain, and tenderness. Systemic reactogenicity events included fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea.
Time Frame: Day 15 through Day 22
Population: The safety population included all participants who received the first dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
Participants
  Pain | 16 | 13
  Tenderness | 20 | 19
  Pruritus | 3 | 0
  Ecchymosis (functional grade) | 1 | 2
  Ecchymosis (measurement grade) | 1 | 2
  Erythema (functional grade) | 3 | 2
  Erythema (measurement grade) | 3 | 2
  Edema/Induration (functional grade) | 2 | 4
  Edema/Induration (measurement grade) | 2 | 3
  Fever | 2 | 2
  Feverishness | 11 | 8
  Fatigue | 16 | 13
  Malaise | 10 | 10
  Myalgia | 10 | 10
  Arthralgia | 5 | 6
  Headache | 14 | 7
  Nausea | 5 | 6

8. Secondary Outcome: Geometric Mean Titer (GMT) and 95% Confidence Interval (CI) of TNA ED50 (Toxin Neutralization Assay 50% Effective Dilution).
Description: Serum for toxin neutralization assay (TNA) was collected at Days 1, 8, 15, 22, 29, 64, 195, and 380. The TNA assay measures the functional ability of antisera containing anti-PA antibodies to specifically protect cells against B. anthracis lethal toxin cytotoxicity. TNA assay results were reported as the reciprocal titer of a serum sample dilution that results in 50% neutralization of lethal toxin cytotoxicity, which is referred to as 50% effective dilution (ED50). To standardize assay results, the results were divided by the ED50 of a serum reference standard, AVR801, and the resulting ratio was reported as a 50% neutralization factor (NF50). Individual results below the lower limit of quantification (LLOQ) for the assay were imputed as 1/2 x LLOQ; the LLOQ for TNA ED50 is 33, so individual results <33 were imputed to 16.5. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1, Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: The modified intent-to-treat (mITT) population included all randomized participants who received the first dose of study vaccine and contributed at least one post-first study vaccination venous blood sample for immunogenicity testing for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
titer
  Day 1 | 16.5 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ. | 17.2 [15.7 to 18.8]
  Day 8 | 16.5 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ. | 22.6 [11.7 to 43.5]
  Day 15 | 21.1 [14.8 to 30.0] | 26.6 [12.9 to 54.7]
  Day 22 | 361.8 [229.2 to 570.9] | 459.9 [273.7 to 772.9]
  Day 29 | 765.9 [572.6 to 1024.6] | 1007.7 [636.6 to 1595.0]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 392.5 [297.4 to 517.9] | 496.5 [312.5 to 788.8]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 97.3 [61.8 to 153.0] | 127.1 [76.2 to 212.2]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 76.3 [47.1 to 123.6] | 103.5 [56.3 to 190.4]

9. Secondary Outcome: Geometric Mean Titer (GMT) and 95% Confidence Interval (CI) of TNA NF50 (Toxin Neutralization Assay 50% Neutralization Factor).
Description: Serum for toxin neutralization assay (TNA) was collected at Days 1, 8, 15, 22, 29, 64, 195, and 380. The TNA assay measures the functional ability of antisera containing anti-PA antibodies to specifically protect cells against B. anthracis lethal toxin cytotoxicity. TNA assay results were reported as the reciprocal titer of a serum sample dilution that results in 50% neutralization of lethal toxin cytotoxicity, which is referred to as 50% effective dilution (ED50). To standardize assay results, the results were divided by the ED50 of a serum reference standard, AVR801, and the resulting ratio was reported as a 50% neutralization factor (NF50). Individual results below the lower limit of quantification (LLOQ) for the assay were imputed as 1/2 x LLOQ; the LLOQ for TNA NF50 is 0.064, so individual results <0.064 were imputed to 0.032. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1, Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
titer
  Day 1 | 0.0320 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ. | 0.0336 [0.0303 to 0.0373]
  Day 8 | 0.0320 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ. | 0.0440 [0.0226 to 0.0855]
  Day 15 | 0.0416 [0.0285 to 0.0605] | 0.0524 [0.0251 to 0.1093]
  Day 22 | 0.7793 [0.4938 to 1.2297] | 0.9394 [0.5559 to 1.5876]
  Day 29 | 1.6211 [1.2078 to 2.1759] | 2.0862 [1.3158 to 3.3077]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 0.8215 [0.6148 to 1.0979] | 1.0668 [0.6823 to 1.6681]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 0.2318 [0.1431 to 0.3753] | 0.3027 [0.1854 to 0.4942]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 0.1885 [0.1182 to 0.3007] | 0.2467 [0.1307 to 0.4654]

10. Secondary Outcome: Geometric Mean Concentration (GMC) and 95% Confidence Interval (CI) of Anti-PA IgG (Anti-protective Antigen Immunoglobulin G)
Description: Serum for anti-PA IgG Enzyme Linked ImmunoSorbent Assay (ELISA) was collected at Days 1, 8, 15, 22, 29, 64, 195, and 380. Individual anti-PA IgG concentrations were reported in µg/mL. Individual results below the lower limit of quantification (LLOQ) for the assay were imputed as 1/2 x LLOQ; the LLOQ for this assay is 9.27 µg/mL, so individual results <9.27 µg/mL were imputed to 4.635 µg/mL. The geometric mean concentration (GMC) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1, Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: concentration (µg/mL)
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
concentration (µg/mL)
  Day 1 | 4.6350 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ. | 4.6350 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ.
  Day 8 | 4.6350 [NA to NA] — 95% CI was not estimable because all values were below the lower limit of quantification (LLOQ) and imputed to 1/2 x LLOQ. | 5.9485 [3.5287 to 10.0275]
  Day 15 | 5.6453 [4.0969 to 7.7789] | 6.4408 [3.5454 to 11.7006]
  Day 22 | 174.8605 [105.2301 to 290.5648] | 99.1012 [62.7645 to 156.4745]
  Day 29 | 342.9604 [253.8561 to 463.3407] | 242.9552 [172.6733 to 341.8433]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 159.5296 [121.2712 to 209.8577] | 126.1505 [85.4090 to 186.3263]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 27.9235 [19.4916 to 40.0029] | 22.3319 [13.3216 to 37.4364]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 14.9907 [9.2110 to 24.3973] | 14.3207 [7.9131 to 25.9170]

11. Secondary Outcome: Percentage and 95% Confidence Interval (CI) of Participants Achieving TNA ED50 (Toxin Neutralization Assay 50% Effective Dilution) Seroconversion.
Description: Serum for toxin neutralization assay (TNA) was collected at Days 1, 8, 15, 22, 29, 64, 195, and 380. The TNA assay measures the functional ability of antisera containing anti-PA antibodies to specifically protect cells against B. anthracis lethal toxin cytotoxicity. TNA assay results were reported as the reciprocal titer of a serum sample dilution that results in 50% neutralization of lethal toxin cytotoxicity, which is referred to as 50% effective dilution (ED50). To standardize assay results, the results were divided by the ED50 of a serum reference standard, AVR801, and the resulting ratio was reported as a 50% neutralization factor (NF50).
  Seroconversion was defined as at least a 4-fold increase over baseline result, or at least a 4-fold increase over the lower limit of quantification (LLOQ) if baseline result is below LLOQ.
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
percentage of participants
  Day 8 | 0 [0 to 16] | 5 [0 to 25]
  Day 15 | 10 [1 to 30] | 5 [0 to 25]
  Day 22 | 86 [64 to 97] | 85 [62 to 97]
  Day 29 | 100 [84 to 100] | 100 [83 to 100]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 100 [83 to 100] | 90 [68 to 99]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 35 [15 to 59] | 35 [15 to 59]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 37 [16 to 62] | 39 [17 to 64]

12. Secondary Outcome: Percentage and 95% Confidence Interval (CI) of Participants Achieving TNA NF50 (Toxin Neutralization Assay 50% Neutralization Factor) Seroconversion.
Description: as for outcome 11
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
percentage of participants
  Day 8 | 0 [0 to 16] | 5 [0 to 25]
  Day 15 | 10 [1 to 30] | 10 [1 to 32]
  Day 22 | 86 [64 to 97] | 85 [62 to 97]
  Day 29 | 100 [84 to 100] | 100 [83 to 100]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 100 [83 to 100] | 100 [83 to 100]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 45 [23 to 68] | 50 [27 to 73]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 47 [24 to 71] | 44 [22 to 69]

13. Secondary Outcome: Percentage and 95% Confidence Interval (CI) of Participants Achieving Anti-PA IgG (Anti-protective Antigen Immunoglobulin G) Seroconversion.
Description: Serum for anti-PA IgG Enzyme Linked ImmunoSorbent Assay (ELISA) was collected at Days 1, 8, 15, 22, 29, 64, 195, and 380. Individual anti-PA IgG concentrations were reported in µg/mL.
  Seroconversion was defined as at least a 4-fold increase over baseline result, or at least a 4-fold increase over the lower limit of quantification (LLOQ) if baseline result is below LLOQ.
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
percentage of participants
  Day 8 | 0 [0 to 16] | 5 [0 to 25]
  Day 15 | 5 [0 to 24] | 5 [0 to 25]
  Day 22 | 86 [64 to 97] | 85 [62 to 97]
  Day 29 | 100 [84 to 100] | 100 [83 to 100]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 100 [83 to 100] | 95 [75 to 100]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 30 [12 to 54] | 25 [9 to 49]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 21 [6 to 46] | 17 [4 to 41]

14. Secondary Outcome: Percentage and 95% Confidence Interval (CI) of Participants Achieving Putative Seroprotection (TNA NF50 = 0.56).
Description: Serum for toxin neutralization assay (TNA) was collected at Days 1, 8, 15, 22, 29, 64, 195, and 380. The TNA assay measures the functional ability of antisera containing anti-PA antibodies to specifically protect cells against B. anthracis lethal toxin cytotoxicity. TNA assay results were reported as the reciprocal titer of a serum sample dilution that results in 50% neutralization of lethal toxin cytotoxicity, which is referred to as 50% effective dilution (ED50). To standardize assay results, the results were divided by the ED50 of a serum reference standard, AVR801, and the resulting ratio was reported as a 50% neutralization factor (NF50).
  Putative seroprotection was defined as TNA NF50 = 0.56.
Time Frame: Day 1, Day 8, Day 15, Day 22, Day 29, Day 64, Day 195, and Day 380
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liquid AV7909 | Lyophilized AV7909
Number analyzed (Participants) | 21 | 20
percentage of participants
  Day 1 | 0 [0 to 16] | 0 [0 to 17]
  Day 8 | 0 [0 to 16] | 5 [0 to 25]
  Day 15 | 5 [0 to 24] | 5 [0 to 25]
  Day 22 | 76 [53 to 92] | 65 [41 to 85]
  Day 29 | 100 [84 to 100] | 85 [62 to 97]
  Day 64: number analyzed (Participants) | 20 | 20
  Day 64 | 65 [41 to 85] | 85 [62 to 97]
  Day 195: number analyzed (Participants) | 20 | 20
  Day 195 | 25 [9 to 49] | 30 [12 to 54]
  Day 380: number analyzed (Participants) | 19 | 18
  Day 380 | 11 [1 to 33] | 33 [13 to 59]

ADVERSE EVENTS:
Time Frame: Reactogenicity was solicited from each study vaccination through Day 8 after vaccination. Unsolicited non-serious adverse events (AEs) were reported from first study vaccination through approximately Day 64. Serious adverse events (SAEs), medically attended adverse events (MAAEs), and adverse events of special interest (AESIs) were collected from first study vaccination through approximately Day 380. Clinical safety laboratory evaluations were performed at approximately Day 29.
Arm/Group | Liquid AV7909 | Lyophilized AV7909
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 21/21 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liquid AV7909 (N=21) | Lyophilized AV7909 (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9) | 8 (9)
Fatigue (General disorders) | 18 (32) | 14 (26)
Injection site erythema (General disorders) | 4 (4) | 3 (4)
Injection site haemorrhage (General disorders) | 3 (3) | 3 (4)
Injection site induration (General disorders) | 4 (4) | 6 (6)
Injection site pain (General disorders) | 21 (41) | 20 (39)
Injection site pruritus (General disorders) | 3 (5) | 2 (2)
Malaise (General disorders) | 14 (20) | 11 (14)
Pyrexia (General disorders) | 12 (16) | 10 (13)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (21) | 10 (16)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 18 (25) | 14 (20)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04660201/Prot_001.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04660201/SAP_002.pdf
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT04660201/ICF_000.pdf